CLINICAL TRIAL: NCT03144895
Title: Arterial Catheterization by Ultrasound: Impact on Success Rates and Complications in Patients Hospitalized in Resuscitation
Brief Title: Arterial Catheterization by Ultrasound
Acronym: ACTIVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2016_843_0014
Record Dates: First submitted 2017-05-02; First posted 2017-05-09 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Ultrasound Therapy; Complications; Intensive Care Unit

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arterial catheter (Other): by anatomical placement alone
  Interventions: Procedure: Laying a radial or femoral arterial catheter
- Placement (Other): of an arterial catheter by ultrasound tracking
  Interventions: Procedure: Laying a radial or femoral arterial catheter

INTERVENTIONS:
Procedure: Laying a radial or femoral arterial catheter — Laying a radial or femoral arterial catheter

SUMMARY:
Monitoring of invasive blood pressure and / or cardiac output of resuscitation patients is required and recommended

DETAILED DESCRIPTION:
Monitoring of invasive blood pressure and / or cardiac output of resuscitation patients is required and recommended. The installation of an arterial catheter in intensive care is very frequent and subject to many complications. These complications are now well recognized in the literature, they are mainly vascular, infectious and thrombotic. They are directly influenced by the number of attempts to puncture and the time taken to perform the gesture. Many measures are taken to reduce the impact such as the choice of the site of installation, the strict aseptic techniques during the installation and the type of catheter used. However, despite these measures, it appears that the incidence of these complications remains high. Compared to anatomical marking, only the technique of laying the ultrasound-guided catheter has shown its effectiveness in reducing these complications. The management in intensive care of increasingly complicated, severe, elderly patients with significant comorbidities increases from year to year. To the knowledge of the investigator, there is no study on the impact of ultrasound arterial catheterization in patients in resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years;
* Hospitalization in resuscitation;
* Necessity of installation of an arterial catheter
* Signed informed consent.
* Affiliation to a social security scheme

Exclusion Criteria:

* Patient under tutorship or curatorship
* Minor Patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2017-03-29 (Actual); Primary Completion 2020-03-28 (Estimated); Study Completion 2020-03-28 (Estimated)

PRIMARY OUTCOMES:
Success rate of arterial or femoral catheter placement | 1 day
  at the first attempted puncture (with only one puncture point on the skin).

CONTACTS AND LOCATIONS:
Overall Officials: Elie ZOGHEIB, PhD, Principal Investigator — CHU AMIENS-PICARDIE
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

REFERENCES:
- [Derived] Flumignan RL, Trevisani VF, Lopes RD, Baptista-Silva JC, Flumignan CD, Nakano LC. Ultrasound guidance for arterial (other than femoral) catheterisation in adults. Cochrane Database Syst Rev. 2021 Oct 12;10(10):CD013585. doi: 10.1002/14651858.CD013585.pub2. PMID 34637140